CLINICAL TRIAL: NCT03051256
Title: Phase 2a Multicenter Randomized Double-Blind Placebo-Controlled Study to Assess the Safety, Tolerability, PK Profile, and Symptom Response of a 7-Day Dosing of REL-1017 as Adjunctive Therapy in the Treatment of Pts Diagnosed With MDD
Brief Title: Safety, Tolerability, PK Profile, and Symptom Response of a 7-Day Dosing With 25 mg or 50 mg Daily of REL-1017 in MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Relmada Therapeutics, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REL-1017-202
Record Dates: First submitted 2017-02-03; First posted 2017-02-13 (Actual); Results first posted 2021-03-17 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant
Keywords: REL-1017; d-Methadone; Methadone; Depression; Refractory Depression; Antidepressant; Adjunctive Treatment; NMDA Receptor Antagonist; Excitatory Amino Acid Antagonist; Glutamate Antagonist
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — D-methadone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- REL-1017 25 mg (Experimental): REL-1017 75 mg of powder in 100 mL of Ocean Spray® Diet Cranberry Juice daily on Day 1, 25 mg of powder in 100 mL Ocean Spray® Diet Cranberry Juice daily on Day 2-7.
  Interventions: Drug: REL-1017
- REL-1017 50 mg (Experimental): REL-1017 100 mg of powder in 100 mL of Ocean Spray® Diet Cranberry Juice daily on Day 1, 50 mg of powder in 100 mL Ocean Spray® Diet Cranberry Juice daily on Day 2-7.
  Interventions: Drug: REL-1017
- Placebo (Placebo Comparator): 100 mL Ocean Spray® Diet Cranberry Juice will be administered as a single oral dose daily for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REL-1017 — REL-1017 will be administered as an oral solution. Patients will continue to take the same, stabilized antidepressant medication that they were taking at screening throughout the course of the study.
  Other Names: d-Methadone
  Arms: REL-1017 25 mg; REL-1017 50 mg
Drug: Placebo — Placebo will be administered as an oral solution. Patients will continue to take the same, stabilized antidepressant medication that they were taking at screening throughout the course of the study.
  Arms: Placebo

SUMMARY:
This a Phase 2a, multicenter, randomized, double-blind, placebo controlled 3 arm study to assess the safety and tolerability of multiple oral doses of REL-1017 25 mg and 50 mg as adjunctive therapy in the treatment of patients diagnosed with major depressive disorder (MDD). The patients will be adults with MDD who are diagnosed with a current MDE who have experienced an inadequate response to 1 to 3 courses of treatment with an antidepressant medication. This population will provide the opportunity to compare the safety and efficacy effects of treatment with an approved antidepressant in conjunction with REL-1017 versus the effects of an antidepressant alone. This study includes in-patient and out-patient periods.

DETAILED DESCRIPTION:
Currently available medications have proven to be useful for the treatment of depression, but also have limitations including low response rates, a significant number of treatment resistant patients, and time-lag for response, which emphasizes a major unmet need for more efficacious and faster-acting antidepressants. Recent studies have demonstrated that ketamine, a non-competitive glutamate-N-methyl-D-Aspartate (NMDA) receptor antagonist, produces rapid onset (2 hours) and long-lasting (7 days) antidepressant actions in treatment resistant patients. This rapid action, by a mechanism completely different from typical monoamine reuptake inhibitors, represents a significant finding in the field of depression.

Racemic methadone, the 50/50 combination of d-methadone and l-methadone, has been in widespread use for decades and has been studied extensively. Methadone is currently approved for use in the management of severe pain, detoxification treatment of opioid addiction, and maintenance treatment of opioid addiction.

The results of a study evaluating the receptor binding profiles of racemic methadone and its stereoisomers suggest that d-methadone does not essentially contribute to the opioid effect of racemic methadone and that it has a 10 times lower affinity for the mu1, mu2, and delta opioid receptors compared to l-methadone. Racemic methadone and its d- and l isomers exhibit similar affinities for the non-competitive binding site of the NMDA receptor and are non-competitive NMDA receptor antagonists.

In the forced swim test, a rodent behavioral model of antidepressant activity, both ketamine and d-methadone at all doses tested significantly decreased the immobility of the rats compared to the vehicle suggesting antidepressant like activity. Neither drug increased spontaneous locomotor activity.

Relmada has conducted 2 clinical studies to identify the dose levels of REL-1017 (d-methadone) that have little to no opioid effects and that are expected to possess NMDA antagonistic properties for the evaluation of oral REL-1017 in the treatment of MDD and neuropathic pain conditions. Initial Phase 1 single ascending dose and multiple ascending dose clinical studies of REL-1017 were designed to evaluate the safety and tolerance of the pure d methadone isomer in healthy opioid-naïve subjects and identify a safe and potentially effective dose range in this population. These studies showed that REL-1017 was safe and well-tolerated at single oral doses up to 150 mg (maximum tolerated dose) and up to 75 mg administered once daily for 10 days in healthy opioid-naïve subjects.

The pre-clinical and previous clinical experience with REL-1017 (d-methadone) provided the basis for the initiation of the present study, which will extend the evaluation of the safety, tolerability, and PK of REL-1017 at 2 doses with repeated administration to depressed patients. Since REL-1017 is proposed for use as adjunctive therapy in the treatment of patients diagnosed with major depressive disorder (MDD), the patients will be male adults with MDD who are diagnosed with a current depressive episode who have experienced an inadequate response to 1 to 3 courses of treatment with an antidepressant medication.

Based on the safety data from Protocol REL-1017-111, single doses of 5 mg, 20 mg, 60 mg, 100 mg, and 150 mg of REL-1017 or placebo were well tolerated. The results of Protocol REL-1017-112 evaluated 10 days of dosing with 25 mg, 50 mg and 75 mg of REL-1017 or placebo, and no impact on safety was observed. In spite of the confirmed dose proportionality, the comparison of concentration and exposure between the 50 mg and 75 mg REL-1017 treatment groups demonstrated only slight differences. Consequently, 25 mg and 50 mg doses were chosen for administration in Protocol REL-1017-202 as single daily doses over a period of 7 days.

Thus, as a single isomer of racemic methadone, d-methadone has been shown to possess NMDA antagonist properties with virtually no opioid activity or ketamine-like toxicities at the expected therapeutic doses.

In this study, adult male patients with MDD who are diagnosed with a current MDE and who have experienced an inadequate response to 1 to 3 courses of treatment with an antidepressant medication will be randomized to study drug in a 1:1:1 ratio. Approximately 15 patients each will receive REL-1017 25 mg, REL-1017 50 mg, or placebo once daily for 7 days. Endpoints include assessments of safety, tolerability, efficacy and pharmacokinetics of REL-1017. Patients will be required to stay in the clinic for 10 days and will then be followed as an outpatient for 12 additional days.

ELIGIBILITY:
Inclusion Criteria:

1. Males between 18 and 65 years of age, inclusive; and females between 18 and 65 years of age, inclusive, who are >1 year postmenopausal.
2. Diagnosed with recurrent MDD as defined by the Diagnostic and Statistical Manual, Fifth Edition (DSM-5), and confirmed by the Mini International Neuropsychiatric Interview, Version 7.0.2 (MINI).
3. Diagnosed with a current MDE lasting 8 weeks to 36 months as defined by the DSM-5 and confirmed by the MINI.
4. Treated with an adequate dosage of a SSRI, SNRI, or bupropion during the current MDE for at least 8 weeks prior to Screening with the same, adequate dosage for the last 4 weeks. Minimum adequate doses are defined in the (ATRQ). The maximum dose allowed for paroxetine is 40 mg QD, for fluoxetine is 60 mg QD, and for sertraline is 200 mg QD.
5. Have experienced an inadequate response to 1 to 3 courses of treatment with an antidepressant medication in the current episode, as defined as <50% improvement with an antidepressant medication at doses listed on the SAFER Interview Criteria: State versus trait; Assessability; Face validity; Ecological validity; and Rule of three Ps (pervasive, persistent, and pathological).
6. Hamilton Depression Rating Scale-17 (HAM-D-17) ≥19 at Screening and Check-in (Day -1).
7. BMI between 18.0 and 35.0 kg/m2, inclusive, and a minimum weight of 50.0 kg.
8. Per the Investigator's judgment, able to meet all study requirements, including the confined/inpatient portion of the study, adherence with both approved ADT and study drug regimen, and completion of all assessments and all scheduled visits.
9. Male patients of reproductive potential must be using and willing to continue using medically acceptable contraception, from Screening and for at least 2 months after the last study drug administration.
10. Must be able to read, speak, and understand English and must provide written informed consent prior to the initiation of any protocol-specific procedures.

Exclusion Criteria:

1. History or presence of clinically significant abnormality as assessed by physical examination, medical history, 12-lead ECG, vital signs, or laboratory values, which in the opinion of the Investigator would jeopardize the safety of the patient or the validity of the study results, including torsades de pointes, any bradyarrhythmias, or uncompensated heart failure.
2. Chronic use of prescribed opioids (i.e., >120 days in a 6-month period) up to 6 months prior to Screening or any recreational use of opioids.
3. Evidence of clinically significant hepatic or renal impairment, including ALT or AST >1.5 x upper limit of normal (ULN), bilirubin >1 x ULN, or endocrine laboratory values (including clinically significant thyroid parameters, i.e., thyroid stimulating hormone [TSH], triiodothyronine [T3], and thyroxine [T4]).
4. History or family history of sudden unexplained death or long QT syndrome (measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle).
5. Any 12-lead ECG with repeated demonstration of QTc ≥450 msec or a QRS interval >120 msec at Screening.
6. History of clinically diagnosed hypotension requiring treatment.
7. History or presence of any condition in which an opioid is contraindicated (e.g., significant respiratory depression, acute or severe bronchial asthma or hypercarbia, bronchitis, or has/is suspected of having paralytic ileus).
8. No more than 3 prescribed doses of an opioid within the 6 months prior to Screening and no use at all within the last month.
9. Use of an antipsychotic, anticonvulsant, or mood stabilizer, regardless of indication, within the 3 months prior to Screening.
10. History of allergy or hypersensitivity to methadone or related drugs (e.g., opioids).
11. Positive test for hepatitis B or HIV. Patients with a positive hepatitis C test may be considered for inclusion with approval from the Medical Monitor.
12. Any current and primary psychiatric disorder, as defined as a condition that is the primary focus of distress and/or treatment, other than MDD.
13. Any lifetime history of bipolar I or II disorder, any psychotic disorder, post-traumatic stress disorder, borderline personality disorder, antisocial personality disorder, obsessive compulsive disorder, eating disorder, intellectual disability, or pervasive developmental disorder.
14. History in the past 12 months of a primary diagnosis of anxiety disorder or panic disorder not related to the current MDE.
15. Current diagnosis of alcohol or substance use disorder, as defined by DSM-5, at Screening or within the 12 months prior to Screening. Patients with the following diagnoses within the past 12 months, however, may be included at the Investigator's discretion: mild alcohol use disorder, mild cannabis use disorder, and any severity tobacco use disorder.
16. A confirmed positive result on the urine drug/alcohol screen at Screening or Check-in. If the urine drug/alcohol screen is positive at Screening, retesting or rescreening may be scheduled with prior approval from the Medical Monitor.
17. Patients who, in the Investigator's judgment, are at significant risk for suicide. A patient with a Columbia-Suicide Severity Rating Scale (C-SSRS) ideation score of 4 or 5 within the last 6 months or any suicide attempt within the past year must be excluded, as should a patient with an ideation score of 4 or 5 or any suicide attempt at the Check-in or Baseline Visit.
18. Patients with a 20% improvement between Screening and Check-in (Day -1) on the HAM-D-17.
19. Patients who did not safely discontinue medications prohibited.
20. Patients receiving new onset psychotherapy (individual, group, marriage, or family therapy) within 2 months prior to Screening or plans to start at any time during participation in the study.
21. Patients who have received electroconvulsive therapy (ECT), repetitive transcranial magnetic stimulation (rTMS), or vagus nerve stimulation (VNS) or who have participated in a ketamine study within the last 6 months.
22. Patients with any clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, chronic pain, or gastrointestinal disorder. Medical conditions that are minor or well-controlled may be permitted if they will not increase the safety risk to the patient or compromise interpretation of the safety or efficacy endpoints.
23. Patients taking fluvoxamine or St. John's Wort.
24. Patients who have participated in a clinical study with an investigational medication in the past 6 months, or who have participated in more than 4 clinical studies with investigational medications in the past 2 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Study Chair — KOL / Advisor
Locations (10):
- United States (10):
  - Woodland International Research Group, Little Rock, Arkansas
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Innovative Clinical Research, Inc, Hialeah, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - St. Louis Clinical Trials, LLC, St Louis, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Midwest Clinical Research Center, Dayton, Ohio
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fava M, Stahl S, Pani L, De Martin S, Pappagallo M, Guidetti C, Alimonti A, Bettini E, Mangano RM, Wessel T, de Somer M, Caron J, Vitolo OV, DiGuglielmo GR, Gilbert A, Mehta H, Kearney M, Mattarei A, Gentilucci M, Folli F, Traversa S, Inturrisi CE, Manfredi PL. REL-1017 (Esmethadone) as Adjunctive Treatment in Patients With Major Depressive Disorder: A Phase 2a Randomized Double-Blind Trial. Am J Psychiatry. 2022 Feb;179(2):122-131. doi: 10.1176/appi.ajp.2021.21020197. Epub 2021 Dec 22. PMID 34933568
- [Result] Guidetti C, Serra G, Pani L, Pappagallo M, Maglio G, Martin S, Mattarei A, Folli F, Manfredi PL, Fava M. Subanalysis of Subjective Cognitive Measures From a Phase 2, Double-Blind, Randomized Trial of REL-1017 in Patients With Major Depressive Disorder. Prim Care Companion CNS Disord. 2023 Feb 14;25(1):22m03267. doi: 10.4088/PCC.22m03267. PMID 36821775
- [Derived] Guidetti C, De Martin S, Serra G, Apicella M, Pani L, Pappagallo M, Mattarei A, Folli F, Manfredi P, Fava M. Effect of Time From Onset of Major Depressive Disorder on the Therapeutic Response to Esmethadone (REL-1017). J Clin Psychiatry. 2024 May 13;85(2):22m14735. doi: 10.4088/JCP.22m14735. PMID 38767937

RESULTS

PARTICIPANT FLOW:
Groups:
- REL-1017 25 mg: Loading dose of REL-1017 75 mg of powder in 100 mL of cranberry juice on Day 1, Maintenance dose of REL-1017 25 mg of powder in 100 mL cranberry juice daily on Days 2-7.
  REL-1017: REL-1017 administered as an oral solution. Patients continued to take the first line stable dose of antidepressant medication.
- REL-1017 50 mg: Loading dose of REL-1017 100 mg of powder in 100 mL of cranberry juice on Day 1, Maintenance dose of REL-1017 50 mg of powder in 100 mL cranberry juice daily on Days 2-7.
  REL-1017: REL-1017 administered as an oral solution. Patients continued to take the first line stable dose of antidepressant medication.
- Placebo: 100 mL cranberry juice was administered as a single oral dose daily for 7 days.
  Placebo: Placebo was administered as an oral solution. Patients continued to take the first line stable dose of antidepressant medication.
Period: Overall Study
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Started | 19 | 21 | 22
Completed (Day 7) | 19 | 21 | 21
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 22 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 22 | 62
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (12.4) | 48.6 (10.9) | 49.7 (11.1) | 49.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 11 | 28
  Male | 11 | 12 | 11 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 13 | 13 | 39
  White | 6 | 7 | 9 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 22 | 62
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.66 (3.33) | 27.66 (5) | 29.02 (4.27) | 28.15 (4.26)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events (AEs) [Safety and Tolerability]
Description: Spontaneously reported or observed AEs will be recorded and reported throughout the study, and AEs will be elicited using a non-leading question at every visit from Screening through the Day 21 assessment.
  An AE was any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and may not necessarily have a causal relationship with the administered treatment. An AE could therefore be any unfavorable and unintended sign (including a clinically significant laboratory abnormality, for example), symptom, or disease temporally associated with the use of a medicinal (investigational) product, regardless of relationship to the medicinal (investigational) product. During the study, an AE could also occur outside the time that the investigational product(s) was given (e.g., during the time from discontinuation of prohibited medications).
Time Frame: 21 days
Population: Safety population: All randomized patients who received any study treatment (REL-1017 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 19 | 21 | 22
Participants
  All-causality TEAEs | 9 | 15 | 12
  All-causality SAEs | 0 | 0 | 0

2. Secondary Outcome: ECG Parameters [Safety]
Description: 12-Lead ECGs will be performed and reported at Screening; at Check In (Day -1); Days 1 through 9; and at Day 14.
Time Frame: Screening, Day -1, Day 1 hour 2, 8, Day 2 hour 2, 8, Day 3-7 hour 2, Day 8, Day 9, and Day 14
Population: Safety population: All randomized patients who received any study treatment (REL-1017 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 19 | 21 | 22
Participants
  Screening: Normal | 14 | 19 | 16
  Screening: Abnormal (not clinically significant) | 5 | 2 | 6
  Screening: Abnormal (clinically significant) | 0 | 0 | 0
  Day -1 (Check-in): Normal | 17 | 19 | 20
  Day -1 (Check-in): Abnormal (not clinically significant) | 2 | 2 | 2
  Day -1 (Check-in): Abnormal (clinically significant) | 0 | 0 | 0
  Day 1, 2 hrs post-dose: Normal | 16 | 18 | 20
  Day 1, 2 hrs post-dose: Abnormal (not clinically significant) | 3 | 3 | 2
  Day 1, 2 hrs post-dose: Abnormal (clinically significant) | 0 | 0 | 0
  Day 1, 8 hrs post-dose: Normal | 15 | 18 | 20
  Day 1, 8 hrs post-dose: Abnormal (not clinically significant) | 4 | 3 | 2
  Day 1, 8 hrs post-dose: Abnormal (clinically significant) | 0 | 0 | 0
  Day 2, 2 hrs post-dose: Normal | 15 | 19 | 20
  Day 2, 2 hrs post-dose: Abnormal (not clinically significant) | 4 | 2 | 2
  Day 2, 2 hrs post-dose: Abnormal (clinically significant) | 0 | 0 | 0
  Day 2, 8 hrs post-dose: number analyzed (Participants) | 19 | 21 | 21
  Day 2, 8 hrs post-dose: Normal | 15 | 19 | 19
  Day 2, 8 hrs post-dose: Abnormal (not clinically significant) | 4 | 2 | 2
  Day 2, 8 hrs post-dose: Abnormal (clinically significant) | 0 | 0 | 0
  Day 3, 2 hrs post-dose: number analyzed (Participants) | 19 | 21 | 21
  Day 3, 2 hrs post-dose: Normal | 14 | 19 | 18
  Day 3, 2 hrs post-dose: Abnormal (not clinically significant) | 5 | 2 | 3
  Day 3, 2 hrs post-dose: Abnormal (clinically significant) | 0 | 0 | 0
  Day 4, 2 hrs post-dose: number analyzed (Participants) | 19 | 21 | 21
  Day 4, 2 hrs post-dose: Normal | 15 | 19 | 19
  Day 4, 2 hrs post-dose: Abnormal (not clinically significant) | 4 | 2 | 2
  Day 4, 2 hrs post-dose: Abnormal (clinically significant) | 0 | 0 | 0
  Day 5, 2 hrs post-dose: number analyzed (Participants) | 19 | 21 | 21
  Day 5, 2 hrs post-dose: Normal | 13 | 19 | 17
  Day 5, 2 hrs post-dose: Abnormal (not clinically significant) | 6 | 2 | 4
  Day 5, 2 hrs post-dose: Abnormal (clinically significant) | 0 | 0 | 0
  Day 6, 2 hrs post-dose: number analyzed (Participants) | 19 | 21 | 21
  Day 6, 2 hrs post-dose: Normal | 15 | 18 | 18
  Day 6, 2 hrs post-dose: Abnormal (not clinically significant) | 4 | 3 | 3
  Day 6, 2 hrs post-dose: Abnormal (clinically significant) | 0 | 0 | 0
  Day 7, 2 hrs post-dose: number analyzed (Participants) | 19 | 21 | 21
  Day 7, 2 hrs post-dose: Normal | 15 | 16 | 19
  Day 7, 2 hrs post-dose: Abnormal (not clinically significant) | 4 | 5 | 2
  Day 7, 2 hrs post-dose: Abnormal (clinically significant) | 0 | 0 | 0
  Day 8: number analyzed (Participants) | 19 | 21 | 21
  Day 8: Normal | 15 | 17 | 19
  Day 8: Abnormal (not clinically significant) | 4 | 4 | 2
  Day 8: Abnormal (clinically significant) | 0 | 0 | 0
  Day 9 (Discharge): number analyzed (Participants) | 19 | 21 | 21
  Day 9 (Discharge): Normal | 14 | 18 | 19
  Day 9 (Discharge): Abnormal (not clinically significant) | 5 | 3 | 2
  Day 9 (Discharge): Abnormal (clinically significant) | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 18 | 19 | 21
  Day 14: Normal | 15 | 17 | 18
  Day 14: Abnormal (not clinically significant) | 3 | 2 | 3
  Day 14: Abnormal (clinically significant) | 0 | 0 | 0

3. Secondary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS) [Safety and Tolerability]
Description: The C-SSRS will be administered and reported at Screening and Check In (Day -1); and at Days 1, 2, 8, 9 and 14.
  The C-SSRS is routinely used to quantify the severity of suicidal ideation and behavior. Both the ideation and behavior subscales are sensitive to change over time.
  The scale identifies behaviors that may be indicative of an individual's intent to commit suicide. This measure contains 6 "yes" or "no" questions in which respondents are asked to indicate whether they have experienced several thoughts or feelings relating to suicide over the past month. Each question addresses a different component of the respondent's suicide ideation severity: (1) Desire to be dead; (2) Suicidal thoughts; (3) Consideration of suicide methods; (4) Formed intent to commit suicide; (5) Completed suicide plan; and (6) Initiated suicide plan. A higher score indicates a higher intensity of suicidal ideation.
Time Frame: Day -1, Day 1, Day 2, Day 8, Day 9 and Day 14
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 100 mL cranberry juice was administered as a single oral dose daily for 7 days.
  Placebo: Placebo will be administered as an oral solution. Patients continued to take the first line stable dose of antidepressant medication.
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 19 | 21 | 22
Participants
  Participants with Suicidal Ideation (Any Score 1-5) : Day -1 (Check-in) | 1 | 0 | 5
  Participants with Suicidal Ideation (Any Score 1-5) : Day 1 (Baseline) | 1 | 0 | 5
  Participants with Suicidal Ideation (Any Score 1-5) : Day 2 | 0 | 0 | 0
  Participants with Suicidal Ideation (Any Score 1-5) : Day 8 | 0 | 1 | 1
  Participants with Suicidal Ideation (Any Score 1-5) : Day 9 (Discharge) | 0 | 1 | 1
  Participants with Suicidal Ideation (Any Score 1-5) : Day 14 | 1 | 1 | 1
  Participants with Suicidal Behavior (any) : Day -1 (Check-in) | 0 | 0 | 0
  Participants with Suicidal Behavior (any) : Day 1 (Baseline) | 0 | 0 | 0
  Participants with Suicidal Behavior (any) : Day 2 | 0 | 0 | 0
  Participants with Suicidal Behavior (any) : Day 8 | 0 | 0 | 0
  Participants with Suicidal Behavior (any) : Day 9 (Discharge) | 0 | 0 | 0
  Participants with Suicidal Behavior (any) : Day 14 | 0 | 0 | 0

4. Secondary Outcome: Montgomery-Asberg Depression Scale (MADRS)
Description: Montgomery-Asberg Depression Scale (MADRS) will be administered and reported on Days 4, 7, and 14.
  The MADRS questionnaire includes questions on the following symptoms: (1) Apparent sadness; (2) Reported sadness; (3) Inner tension; (4) Reduced sleep; (5) Reduced appetite; (6) Concentration difficulties; (7) Lassitude; (8) Inability to feel; (9) Pessimistic thoughts; (10) Suicidal thoughts.
  A higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60 with scores above 34 indicating severe depression. In Study REL-1017-202, the MADRS was administered using the Structured Interview Guide for the MADRS (SIGMA).
  A negative change from baseline indicates improvement.
Time Frame: Change from Baseline to Day 7
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 19 | 21 | 21
score on a scale | -17.4 (2.5) | -15.9 (2.4) | -8.7 (2.3)
Statistical Analysis 1: Comparison: REL-1017 25 mg vs Placebo; Test type: Superiority; p < 0.0122, Mixed Models Analysis
Statistical Analysis 2: Comparison: REL-1017 50 mg vs Placebo; Test type: Superiority; p < 0.0308, Mixed Models Analysis

5. Secondary Outcome: Montgomery-Asberg Depression Scale (MADRS)
Description: as for outcome 4
Time Frame: Change from Baseline to Day 14
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 16 | 18 | 20
score on a scale | -16.8 (2.7) | -17.8 (2.6) | -7.4 (2.4)
Statistical Analysis 1: Comparison: REL-1017 25 mg vs Placebo; Test type: Superiority; p < 0.0103, Mixed Models Analysis
Statistical Analysis 2: Comparison: REL-1017 50 mg; Test type: Superiority; p < 0.0039, Mixed Models Analysis

6. Secondary Outcome: Symptoms of Depression Questionnaire (SDQ)
Description: Symptoms of Depression Questionnaire (SDQ) will be administered and reported on Days 4, 7, and 14.
  The SDQ is a 44-item, self-report scale designed to measure the severity of symptoms across several subtypes of depression. The SDQ was developed to more fully capture the heterogeneity of symptom presentations of depressive disorders than current, widely used scales for MDD. The SDQ includes items that inquire about an extensive number of depressive symptoms beyond the ones included in other commonly used scales. The 44 SDQ items are rated on a 6-point scale. The total score is the sum of 44 items and can range from 44 to 264. A negative change from baseline indicates improvement.
  1 = Better than Normal; 2= Normal; 3= Minimally Sad; 4= Moderately Sad; 5= Markedly Sad; 6= Extremely Sad
Time Frame: Change from Baseline to Day 7
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 19 | 21 | 21
score on a scale | -52.4 (7.1) | -52.9 (6.6) | -37.9 (6.4)
Statistical Analysis 1: Comparison: REL-1017 25 mg vs Placebo; Test type: Superiority; p = 0.1237, Mixed Models Analysis
Statistical Analysis 2: Comparison: REL-1017 50 mg vs Placebo; Test type: Superiority; p = 0.1017, Mixed Models Analysis

7. Secondary Outcome: Symptoms of Depression Questionnaire (SDQ)
Description: as for outcome 6
Time Frame: Change from Baseline to Day 14
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 16 | 18 | 20
score on a scale | -55.0 (6.4) | -58.6 (6.0) | -31.8 (5.6)
Statistical Analysis 1: Comparison: REL-1017 25 mg vs Placebo; Test type: Superiority; p < 0.0066, Mixed Models Analysis
Statistical Analysis 2: Comparison: REL-1017 50 mg vs Placebo; Test type: Superiority; p < 0.0014, Mixed Models Analysis

8. Secondary Outcome: Clinical Global Impressions of Severity (CGI-S)
Description: Clinical Global Impressions of Severity (CGI-S) will be administered and reported on Days 4, 7, and 14.
  The CGI-S is a standard method used in clinical studies to quantify and track patient progress and treatment response over time. The scale is composed of 7 ratings: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. The score ranges from 1 to 7, and a lower CGI-S score indicates lower levels of depression.
Time Frame: Change from Baseline to Day 7
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 19 | 21 | 21
score on a scale | -1.7 (0.3) | -1.7 (0.3) | -0.8 (0.3)
Statistical Analysis 1: Comparison: REL-1017 25 mg vs Placebo; Test type: Superiority; p < 0.0245, Mixed Models Analysis
Statistical Analysis 2: Comparison: REL-1017 50 mg vs Placebo; Test type: Superiority; p < 0.0253, Mixed Models Analysis

9. Secondary Outcome: Clinical Global Impressions of Severity (CGI-S)
Description: as for outcome 8
Time Frame: Change from Baseline to Day 14
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 16 | 18 | 20
score on a scale | -1.6 (0.3) | -2.0 (0.3) | -0.7 (0.3)
Statistical Analysis 1: Comparison: REL-1017 25 mg vs Placebo; Test type: Superiority; p < 0.0454, Mixed Models Analysis
Statistical Analysis 2: Comparison: REL-1017 50 mg vs Placebo; Test type: Superiority; p < 0.0043, Mixed Models Analysis

10. Secondary Outcome: Clinical Global Impressions of Improvement (CGI-I)
Description: Clinical Global Impressions of Improvement (CGI-I) will be administered and reported at Days 4, 7 and 14.
  The CGI-I is a standard method used in clinical studies to quantify and track patient change over time. The scale is composed of 7 ratings: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; and 7 = very much worse. The score ranges from 1 to 7, and a lower CGI-I score indicates greater improvement in symptoms.
Time Frame: Change from Baseline to Day 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 19 | 21 | 21
score on a scale | 2.4 (0.2) | 2.3 (0.2) | 3.2 (0.2)
Statistical Analysis 1: Comparison: REL-1017 25 mg vs Placebo; Test type: Superiority; p = 0.0177, Mixed Models Analysis
Statistical Analysis 2: Comparison: REL-1017 50 mg vs Placebo; Test type: Superiority; p = 0.0072, Mixed Models Analysis

11. Secondary Outcome: Clinical Global Impressions of Improvement (CGI-I)
Description: as for outcome 10
Time Frame: Change from Baseline to Day 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
Number analyzed (Participants) | 16 | 18 | 20
score on a scale | 2.6 (0.3) | 2.3 (0.3) | 3.3 (0.3)
Statistical Analysis 1: Comparison: REL-1017 25 mg vs Placebo; Test type: Superiority; p = 0.0895, Mixed Models Analysis
Statistical Analysis 2: Comparison: REL-1017 50 mg vs Placebo; Test type: Superiority; p = 0.0109, Mixed Models Analysis

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) [Pharmacokinetic]
Description: The pharmacokinetic parameters of REL-1017 25 mg and 50 mg will be evaluated on Day 1 through Day 7, Day 8, Day 9, and Day 14 where the data allow.
Time Frame: Day 1 (hour -1, 1, 2, 4, 6, 8, 12, and 24)
Population: Pharmacokinetic population: All patients who received REL-1017, with at least 1 post-dose blood draw to determine plasma concentration of d-methadone.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | REL-1017 25 mg | REL-1017 50 mg
Number analyzed (Participants) | 16 | 21
ng/mL | 254.5 (60.864) | 343.9 (112.36)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Until the Dosing Interval of 24 Hours (AUCtau) [Pharmacokinetic]
Description: as for outcome 12
Time Frame: Day 1 (hour -1, 1, 2, 4, 6, 8, 12, and 24)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | REL-1017 25 mg | REL-1017 50 mg
Number analyzed (Participants) | 16 | 20
h*ng/mL | 3533 (1082.2) | 4531 (1344.7)

14. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) [Pharmacokinetic]
Description: as for outcome 12
Time Frame: Day 1 (hour -1, 1, 2, 4, 6, 8, 12, and 24)
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | REL-1017 25 mg | REL-1017 50 mg
Number analyzed (Participants) | 16 | 21
hours | 1.917 [0.950 to 6.00] | 2.250 [1.00 to 6.02]

15. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) [Pharmacokinetic]
Description: as for outcome 12
Time Frame: Day 1 (hour -1, 1, 2, 4, 6, 8, 12, and 24)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | REL-1017 25 mg | REL-1017 50 mg
Number analyzed (Participants) | 11 | 15
h*ng/mL | 7114 (2685.2) | 10190 (5627.6)

16. Secondary Outcome: Apparent Terminal Elimination Half-life (t½) [Pharmacokinetic]
Description: as for outcome 12
Time Frame: Day 1 (hour -1, 1, 2, 4, 6, 8, 12, and 24) and Day 7 (hour 24, 48, and 168 post last dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: h
Arm/Group | REL-1017 25 mg | REL-1017 50 mg
Number analyzed (Participants) | 16 | 20
h
  Day 1 | 30.60 (18.739) | 31.74 (18.888)
  Day 7: number analyzed (Participants) | 9 | 7
  Day 7 | 43.88 (11.621) | 38.16 (3.9399)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | REL-1017 25 mg | REL-1017 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 9/19 | 15/21 | 12/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REL-1017 25 mg (N=19) | REL-1017 50 mg (N=21) | Placebo (N=22)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Weight Decrease (Investigations) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritius (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Increases (Investigations) | 0 (0) | 1 (1) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Application Site Erosion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling of Relaxation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor requests an opportunity to review any proposed publication prior to public release to ensure against inadvertent release of confidential information or unprotected inventions. Sponsor has 12 months from the completion or termination of the trial to publish a joint manuscript with all participating sites.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT03051256/Prot_SAP_000.pdf